CLINICAL TRIAL: NCT01511991
Title: Sevoflurane's Effect on Tissue Doppler Profiles of Lateral Mitral Annulus During Cardiac Surgery
Brief Title: Sevoflurane's Effect on Mitral Valve Annular Velocity in Cardiac Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: KUH1160037
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Valvular Heart Disease
Keywords: cardiac surgery; sevoflurane; tissue Doppler
MeSH Terms: conditions — Heart Valve Diseases | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sevoflurane (Experimental): 10 min exposure to sevoflurane 1.0, 2.0 and 3.0 inspiratory vol% at sevoflurane dosage titration
  Interventions: Drug: Sevoflurane dosage titration

INTERVENTIONS:
Drug: Sevoflurane dosage titration — comparisons of the effect of the 10 min-inhalation of each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3)
  Other Names: sevorane

SUMMARY:
The purpose of this study is to determine sevoflurane's dose-dependent effect on left ventricular (LV) function in cardiac surgery. The change of tissue Doppler imaging (TDI) of lateral mitral valve annular velocity at three different sevoflurane concentrations would be analyzed by using intraoperative transesophageal echocardiography (TEE)in cardiac surgery patients.

DETAILED DESCRIPTION:
Following data would be determined after 10 min-exposure to each dosage of sevoflurane with 1.0, 2.0 and 3.0 inspired vol% (T1, T2 and T3, respectively) during remifentanil-based anesthesia (1.0 mcg/kg/min) for cardiac surgery (n=14):

1. TDI of lateral mitral annulus at systole (S'), early filling (E') and atrial contraction (A')
2. transmitral flow Doppler at early filling (E), atrial contraction (A), deceleration time;
3. LV-ejection fraction (EF)
4. bispectral index (BIS)
5. phenylephrine-infusion rate
6. other pressure derived hemodynamic parameters:heart rate; systolic, diastolic, and mean blood pressures; systolic, diastolic, and mean pulmonary artery pressures; central venous pressure (CVP), pulmonary capillary wedge pressure (PCWP), mixed venous O2 saturation (SvO2), cardiac index (CI) and stroke volume index (SVI)

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery

Exclusion Criteria:

* low ejection fraction < 50% in preoperative transthoracic echocardiography
* atrial fibrillation
* pacemaker
* pericardial and infiltrative myocardial disease
* mitral annular calcification, surgical rings, prosthetic mitral valves
* lateral left ventricular regional wall motion abnormality
* esophageal spasm,stricture, laceration, perforation, and diverticulum
* diaphragmatic hernia,
* history of extensive radiation to the mediastinum
* upper gastrointestinal bleeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Peak mitral annular velocity during systole (S') | after 10 min exposure to sevoflurane 1.0 vol%, 2.0 vol% and 3.0 vol%
  By using pulsed Doppler with the sample volume positioned at the lateral MV ring in the midesophageal 4-chamber view, S' would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)
Peak mitral annular velocity during early filling (E') | after 10 min exposure to sevoflurane of 1.0 vol%, 2.0 vol% and 3.0 vol%
  By using pulsed Doppler with the sample volume positioned at the lateral MV ring in the midesophageal 4-chamber view, E' would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)
peak mitral annular velocity during atrial contraction(A') | after 10 min exposure to sevoflurane 1.0 vol%, 2.0 vol% and 3.0 vol%
  By using pulsed Doppler with the sample volume positioned at the lateral MV ring in the midesophageal 4-chamber view, A' would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)

SECONDARY OUTCOMES:
ejection fraction (EF) | after 10 min exposure to sevoflrane 1.0vol%, 2.0 vol% and 3.0 vol%
  By using modified Simpson technique in the midesophageal 4-chamber view, EF would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)
bispectral index (BIS) | after 10 min exposure to sevoflurane 1.0 vol%, 2.0 vol% and 3.0 vol%
  BIS would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)
peak velocity of mitral inflow during early relaxation (E) | after 10 min exposure to sevoflurane 1.0 vol%, 2.0 vol% and 3.0 vol%
  By using pulsed Doppler with the sample volume positioned at the lMV opening in the midesophageal 4-chamber view, S' would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)
peak velocity of mitral inflow during atrial contraction (A) | after 10 min exposure to sevoflurane 1.0 vol%, 2.0 vol% and 3.0 vol%
  By using pulsed Doppler with the sample volume positioned at the tip of MV oeneing in the midesophageal 4-chamber view, "A" would be determined just after the 10 min-exposure to each concentration of sevoflurane, 1.0 inspired vol%, 2.0 inspired vol% and 3.0 inspired vol% (T1, T2 and T3, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Bruch C, Gradaus R, Gunia S, Breithardt G, Wichter T. Doppler tissue analysis of mitral annular velocities: evidence for systolic abnormalities in patients with diastolic heart failure. J Am Soc Echocardiogr. 2003 Oct;16(10):1031-6. doi: 10.1016/S0894-7317(03)00634-5. PMID 14566295
- [Background] Waggoner AD, Bierig SM. Tissue Doppler imaging: a useful echocardiographic method for the cardiac sonographer to assess systolic and diastolic ventricular function. J Am Soc Echocardiogr. 2001 Dec;14(12):1143-52. doi: 10.1067/mje.2001.115391. PMID 11734780